CLINICAL TRIAL: NCT01147029
Title: A Cancer Research UK Phase I Trial of 4-(N-(S-Glutathionylacetyl) Amino) Phenylarsenoxide (GSAO) Given as Daily Intravenous Infusions on Days 1-5 and 8-12 of a 21-Day Cycle, to Patients With Advanced Solid Tumors
Brief Title: GSAO in Treating Patients With Advanced Solid Tumors That Have Not Responded to Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000675271; CRUK-PH1-109; EUDRACT-2006-002326-34; CTA-21106-0222-001
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 4-(N-(S-glutathionylacetyl)amino)phenylarsenoxide

INTERVENTIONS:
Drug: angiogenesis inhibitor GSAO
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: dynamic contrast-enhanced magnetic resonance imaging

SUMMARY:
RATIONALE: GSAO may stop the growth of solid tumors by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of GSAO in treating patients with advanced solid tumors that have not responded to therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose and recommended phase II dose of angiogenesis inhibitor GSAO in patients with advanced, refractory solid tumors.
* To assess the safety and toxicity profile and dose-limiting toxicity of this drug in these patients.

Secondary

* To determine the pharmacokinetics of this drug in these patients.
* To determine the pharmacodynamics of this drug in these patients.
* To determine possible anti-tumor activity in patients treatment with this drug.

Tertiary

* To further determine the pharmacodynamics of this drug in these patients.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive angiogenesis inhibitor GSAO IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients showing clinical benefit (i.e., stable disease, partial response, or complete response) may receive 6 additional courses of treatment. Patients receive angiogenesis inhibitor GSAO IV over 1 hour on day -7 to obtain pharmacokinetics information of a single IV dose of the drug.

Patients also undergo dynamic contrast-enhanced magnetic-resonance imaging (DCE-MRI) prior to, during, and after study to determine blood flow parameters.

Blood samples are collected periodically for pharmacokinetic, pharmacodynamic, and biomarker studies.

After completion of study treatment, patients are followed up for 28 days and then once a month thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor

  * Refractory to conventional treatment or for which no conventional therapy exists
* Disease assessable by DCE-MRI and should be of a size that can be adequately assessed by these techniques
* No known primary brain tumors or brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100 x 10^9/L
* Neutrophil count ≥ 1.5 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Creatinine clearance ≥ 50 mL/min (uncorrected value)
* Serum potassium and magnesium normal
* No proteinuria > grade 1 either on 24-hour urine or on 2 consecutive dipsticks taken no less than 1 week apart
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 4 weeks prior to, during, and for 6 months after completion of study therapy
* Not at high medical risk due to non-malignant systemic disease, including active uncontrolled infection
* No serologically positive hepatitis B, hepatitis C, or HIV
* No concurrent congestive heart failure or prior NYHA class III-IV cardiac disease
* None of the following medical conditions:

  * Angina (stable or severe, even if well controlled on medication)
  * Myocardial infarction in the past 2 months by ECG
  * Congestive cardiac failure
  * Arrhythmias, including any condition associated with QTc prolongation (e.g., Lange-Neilson syndrome or Romano Ward syndrome)
  * Evidence of ischemia
  * QTc > 480 msec
  * Other clinically significant abnormalities
* No uncontrolled hypertension (defined as BP consistently greater than 160/100 mm Hg irrespective of medication)
* No other condition that, in the opinion of the investigator, would not make the patient a good candidate for this clinical trial
* No pacemakers
* No metal fragments in the eyes or shrapnel or bullet injuries

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior treatments (except for alopecia or certain grade 1 toxicities which, in the opinion of the investigator and Cancer Research UK, should not exclude the patient)
* At least 4 weeks since prior radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy, or chemotherapy (6 weeks for nitrosoureas and mitomycin C)
* At least 1 week since prior and no concurrent shellfish
* At least 6 weeks since prior major surgery (including thoracic and/or abdominal surgery) and recovered
* Concurrent luteinizing-hormone releasing-hormone (LHRH) analogues allowed for patients with castration-refractory prostate cancer provided the prostate-specific antigen level is rising
* No prior heart or brain surgery
* No concurrent drug known to prolong the QTc interval
* No concurrent warfarin (1 mg for maintenance of a Hickman line is acceptable) or heparin (flushing of arterial lines, if necessary, is acceptable)
* No concurrent naproxen (other NSAIDs are acceptable)
* No concurrent prophylactic use of antiemetics during the first treatment

  * Domperidone and lorazepam must not be used as antiemetics
* No other concurrent anticancer therapy or investigational drugs

  * Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity
Causality of each adverse event and grading severity according to NCI CTCAE Version 3.0

SECONDARY OUTCOMES:
Relationship between pharmacokinetics and toxicity and/or markers of efficacy
Changes in microvascular function using DCE-MRI
Plasma and tumor levels of angiogenic factors and apoptosis markers
Response (stable disease, partial response, or complete response) as determined by RECIST criteria
Circulating endothelial cells and circulating endothelial progenitor cells as a marker of inhibition of angiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Christie Hospital, Manchester, England
  - Churchill Hospital, Oxford, England